CLINICAL TRIAL: NCT03881722
Title: Effect of Magnesium Alginate in Infants With Gastroesophageal Reflux.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, Researcher, Policlinico Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALGNEO1
Record Dates: First submitted 2018-02-17; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomized controlled cross-over trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thickened formula (Active Comparator)
  Interventions: Dietary Supplement: Mg alginate
- Mg alginate (Experimental)
  Interventions: Dietary Supplement: Mg alginate

INTERVENTIONS:
Dietary Supplement: Mg alginate — Mg alginate after feedings

SUMMARY:
Recurrent regurgitation stress the infants and their parents and often results in an inappropirate use of PPI prescription in infancy. The aim of this study is to evaluate the efficacy of Mg alginate in infants with symptoms of gastroesophageal reflux.

ELIGIBILITY:
Inclusion Criteria:

* symptoms suggestive of GER, evaluated through a validated questionnaire (Infant Gastroesophageal Reflux Questionnaire Revised: I-GERQ-R > 16)
* informed consent signed

Exclusion Criteria:

* congenital or chronic diseases
* use of anti acid drugs

Ages: 3 Weeks to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Infant Gastro-Esophageal Reflux Questionnaire Revised | through study completion, an average of 1 month
  12-item validated questionnaire called Infant Gastro-Esophageal Reflux Questionnaire Revised (I-GERQ-R) which include different questions about regurgitation, crying, feeding and respiratory problems

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Of Obstetrics and Neonatology - Section of Neonatology University of Bari Policlinico Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: No